CLINICAL TRIAL: NCT02061826
Title: Establishment of Drug-induced Liver Injury Databases and Application of Circulating miRNA
Brief Title: Establishment of Drug-induced Liver Injury Databases and Application of Circulating microRNA(miRNA)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wen Xie, head of department, Beijing Ditan Hospital
Other Study IDs: Ditan-2014-01
Record Dates: First submitted 2014-01-26; First posted 2014-02-13 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Drug-induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood, serum,plasma,PBMC
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to establish drug-induced liver injury databases in China, make criteria for Chinese drug-induced liver injury patients and evaluate the application of certain circulating miRNA in diagnosis or treatment of drug-induced liver injury.

DETAILED DESCRIPTION:
Firstly, this study collects some retrospective data. Analyse these data and establish certain unique diagnostic criteria for Chinese. Then collect prospective data and validate the criteria. Otherwise,collect blood sample or other sample of the patients and study certain miRNA in diagnosis or treatment of drug-induced liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 18 to 70 years
* Women in child-bearing period taking some contraception measures
* Patients with onset of acute liver injury attributed to antituberculosis drugs or antineoplastic drugs, Roussel Uclaf Causality Assessment Method（RUCAM ） score≥6
* Written informed consent can be obtained, some patients agree with liver biopsy

Exclusion Criteria:

* Viral hepatitis
* Alcoholic liver disease or non-alcoholic liver disease
* Wilson's disease or other inherited metabolic liver diseases
* Auto-immune liver diseases
* Any dysfunction of liver
* Malnutrition
* Chronic diseases such as HIV,severe heart diseases, severe brain diseases or chronic kidney diseases
* Patients who can not complete follow-ups on time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample and primary care clinic
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
histological features of drug-induced liver injury obtained by liver biopsy | within six months of the DILI onset date
  Liver biopsy is the main method
clinical features of drug-induced liver injury assessed by serum parameters of liver function | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  serum parameters of liver function is the focus

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xie, master, Study Director — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Beijing, China